CLINICAL TRIAL: NCT05763459
Title: A Phase 1 Study to Evaluate the Drug-Drug Interaction Between ABBV-CLS-7262, Rosuvastatin, and Digoxin Following Multiple Doses of ABBV-CLS-7262
Brief Title: A Phase 1 Study of ABBV-CLS-7262, Rosuvastatin, and Digoxin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calico Life Sciences LLC (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M24-192
Record Dates: First submitted 2023-02-27; First posted 2023-03-10 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Digoxin; Rosuvastatin; Molecular Mechanisms of Pharmacological Action; Physiological effects of drugs

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABBV-CLS-7262 (Experimental): ABBV-CLS-7262 + Digoxin + Rosuvastatin
  Interventions: Drug: ABBV-CLS-7262

INTERVENTIONS:
Drug: ABBV-CLS-7262 — Drug: ABBV-CLS-7262 Drug: Digoxin Drug: Rosuvastatin

SUMMARY:
This study follows an open-label, single arm design with two periods with rosuvastatin, digoxin and ABBV-CLS-7262

DETAILED DESCRIPTION:
Period 1: One single dose of rosuvastatin and one single dose of digoxin on Day 1.

Period 2: Multiple doses of ABBV-CLS-7262 once daily from Day 1 to Day 8. On Day 5, one single dose of rosuvastatin and one single dose of digoxin with the dose of ABBV-CLS-7262 on that day.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers in general good health
* Must voluntarily sign and date an informed consent, approved by an independent ethics committee (IEC)/institutional review board (IRB), prior to the initiation of any screening or study-specific procedures
* Individuals between 18 and 65 years of age inclusive at the time of screening
* BMI is ≥ 18.0 to ≤ 32.0 kg/m2
* All male subjects who are sexually active and not surgically sterilized must agree to use an acceptable contraceptive method. Additionally, male subjects must agree to not donate sperm during the study until 30 days after the final dose of study drug
* All female subjects who are sexually active and of childbearing potential must agree to use a highly effective contraceptive method. Additionally, female subjects must agree to not donate eggs during the study and for 30 days after the final dose of study drug.

Exclusion Criteria:

* Subject who, in the opinion of the investigator, is incapable of completing study-required visits and procedures
* Pregnant or breastfeeding.
* Treatment with any other investigational treatment within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Rosuvastatin | Two Weeks
  Area under the Curve (AUC)
Pharmacokinetics of Digoxin | Two Weeks
  Area under the Curve (AUC)

SECONDARY OUTCOMES:
Safety and Tolerability | Two Weeks
  Number of patients with treatment-related adverse events as assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- AbbVie Clinical Pharmacology Research Unit (ACPRU), Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No